CLINICAL TRIAL: NCT00001045
Title: A Double-Blinded, Randomized Trial Comparing Zidovudine (AZT) Versus AZT Plus Didanosine (ddI) Versus AZT Plus ddI Plus Nevirapine in Asymptomatic Patients on AZT Monotherapy Who Develop a Mutation at Codon 215 of HIV Reverse Transcriptase in Serum/Plasma Viral RNA
Brief Title: Comparison of Three Anti-HIV Drug Combinations in HIV-Infected Patients With No Symptoms of the Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry); Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 244; 11221 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Zidovudine; Nevirapine
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine; Zidovudine; Didanosine

INTERVENTIONS:
Drug: Nevirapine
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
To validate that the alteration of codon 215 of reverse transcriptase in plasma virus precedes the increase in viral burden as measured in the peripheral blood and the decline in CD4 count that have been observed in association with clinical failure on zidovudine (AZT). To determine whether alternative regimens of antiretroviral agents alter the course of viral burden as measured in the peripheral blood and CD4 changes in patients with HIV infection. To obtain further data on the safety and immunologic and virologic response to AZT/didanosine/nevirapine.

Of the HIV-1 mutations reported to be associated with zidovudine resistance, the mutation at codon 215 of the reverse transcriptase gene is the most commonly occurring and has the greatest impact on susceptibility. When this mutation appears, a change in drugs may prevent further immunologic and virologic deterioration.

DETAILED DESCRIPTION:
Of the HIV-1 mutations reported to be associated with zidovudine resistance, the mutation at codon 215 of the reverse transcriptase gene is the most commonly occurring and has the greatest impact on susceptibility. When this mutation appears, a change in drugs may prevent further immunologic and virologic deterioration.

Initially, all patients receive AZT alone. After detection of a 215 mutation in plasma RNA, patients are randomized to one of three treatment arms: AZT alone, AZT plus ddI, or AZT/ddI plus nevirapine. Patients are followed every 8 weeks and receive treatment for up to 4 years.

AS PER AMENDMENT 5/9/96: All AZT monotherapy options have been eliminated. Patients will be randomized to either Arm II or Arm III, regardless of their codon 215 status. All patients who were randomized to Arm I following a mutation at codon 215 will be rerandomized to Arm II or Arm III. All patients who were randomized to either Arm II or Arm III following a mutation at codon 215 will remain on their initial randomized assignment.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Chemoprophylaxis for Pneumocystis carinii pneumonia.
* Antibiotics, antifungals, and antiviral medications, as clinically indicated.
* Regularly prescribed medication such as antipyretics, analgesics, allergy medications, antidepressants, sleep medications, oral contraceptives, or any other medications deemed appropriate by the primary care provider.

Concurrent Treatment:

Allowed:

* Limited localized radiation therapy to the skin.

Prior Medication: Required:

* AZT (minimum 300 mg/day) for at least 1 month (uninterrupted) but no more than 2 years immediately prior to study entry.

Patients must have:

* Asymptomatic HIV infection.
* CD4 count 300-600 cells/mm3.
* No plasma/serum PCR for codon 215 mutation at screening.
* Prior AZT monotherapy.

NOTE:

* All Department of Defense (DOD)-eligible patients must be at least 18 years of age. Enrollment of women is encouraged.

AS PER AMENDMENT 04/03/95:

* DOD female patients must have a negative pregnancy test within 48 hours prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Symptomatic grade 2 or worse peripheral neuropathy.
* Unable to swallow capsules and tablets.
* Other medical condition that contraindicates study participation.

Concurrent Medication:

Excluded:

* Systemic cytotoxic chemotherapy.
* Biologic response modifiers (such as interferon, ampligen, or PEG-IL2).
* Anti-HIV agents other than study drugs.
* Other investigational agents.
* Foscarnet unless clinically indicated for unresponsive herpes virus infection.
* Chronic antacid or H-2 blocker use.
* Rifampin or rifamycin class agents.
* Antibiotics containing clavulanic acid.

Concurrent Treatment:

Excluded:

* Radiation therapy other than limited localized therapy to skin.

Patients with the following prior condition are excluded:

* History of pancreatitis.

Prior Medication:

Excluded:

* Prior therapy with nucleoside or non-nucleoside antiretroviral agents other than AZT.
* Immune modulating therapies (e.g., IFN-alpha, gp160) within 60 days prior to screening.

Prior Treatment:

Excluded:

* Blood transfusion within the preceding 2 weeks.

Illicit drug or alcohol abuse.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Study Completion 1998-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merigan TC, Study Chair; Mayers DL, Study Chair
Locations (59):
- United States (57):
  - UCLA CARE Ctr, Los Angeles, California
  - Stanford at Kaiser / Kaiser Permanente Med Ctr, San Francisco, California
  - Santa Clara Valley Med Ctr / AIDS Community Rsch Consortium, San Jose, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Children's Hosp of Washington DC, Washington D.C., District of Columbia
  - George Washington Univ / Hershey Med Ctr, Washington D.C., District of Columbia
  - Walter Reed Army Med Ctr, Washington D.C., District of Columbia
  - Emory Univ Hosp / Pediatrics, Atlanta, Georgia
  - Emory Hemo Comp Evaluation Clinic / East TN Comp Hemo Ctr, Atlanta, Georgia
  - Queens Med Ctr, Honolulu, Hawaii
  - Univ of Hawaii, Honolulu, Hawaii
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Univ of Iowa Hosp and Clinic, Iowa City, Iowa
  - State of MD Div of Corrections / Johns Hopkins Univ Hosp, Baltimore, Maryland
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Natl Naval Med Ctr, Bethesda, Maryland
  - Fitzsimmons Army Med Ctr, Rockville, Maryland
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Hennepin County Med Clinic, Minneapolis, Minnesota
  - Univ of Minnesota, Minneapolis, Minnesota
  - St Paul Ramsey Med Ctr, Saint Paul, Minnesota
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - Adirondack Med Ctr at Saranac Lake, Albany, New York
  - Albany Med College / Division of HIV Medicine A158, Albany, New York
  - Mid - Hudson Care Ctr, Albany, New York
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - SUNY / State Univ of New York, Syracuse, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Comprehensive Health Care Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Family Health Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Jack Weiler Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Med Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Med Ctr Adolescent AIDS Program, The Bronx, New York
  - North Central Bronx Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Carolinas Med Ctr, Charlotte, North Carolina
  - Wake County Dept of Health, Raleigh, North Carolina
  - Case Western Reserve Univ, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Med College of Ohio, Toledo, Ohio
  - Milton S Hershey Med Ctr, Hershey, Pennsylvania
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson Univ Hosp, Philadelphia, Pennsylvania
  - Univ of Tennessee / E Tennessee Comprehensive Hemophilia Ctr, Knoxville, Tennessee
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Univ of Texas Galveston, Galveston, Texas
  - Wilford Hall Med Ctr, Lackland Air Force Base, Texas
  - Brooke Army Med Ctr, San Antonio, Texas
- Puerto Rico (2):
  - Ramon Ruiz Arnau Univ Hosp / Pediatrics, Bayamón
  - San Juan City Hosp, San Juan

REFERENCES:
- [Background] Slade DE, Vavro CL, Stapleton JT, Swack N, StClair MH. A novel mutation at codon 215 of HIV RT. Int Conf AIDS. 1993 Jun 6-11;9(1):239 (abstract no PO-A26-0625)
- [Background] Mayers D, Merigan T, Gilbert P. T215Y/F mutation associated with zidovudine (ZDV) resistance leads to poor response to ZDV+ddI or ZDV+ddI+NVP: ACTG244/RV79. Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:91 (abstract no 129)
- [Background] Holodniy M, Katzenstein D, Mole L, Winters M, Merigan T. Human immunodeficiency virus reverse transcriptase codon 215 mutations diminish virologic response to didanosine-zidovudine therapy in subjects with non-syncytium-inducing phenotype. J Infect Dis. 1996 Oct;174(4):854-7. doi: 10.1093/infdis/174.4.854. PMID 8843229